CLINICAL TRIAL: NCT00004380
Title: Phase II Study of Recombinant Relaxin for Progressive Systemic Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Stanford University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: 199/12015; SUMC-37488
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-07

CONDITIONS: Systemic Sclerosis
Keywords: arthritis & connective tissue diseases; rare disease; systemic sclerosis
MeSH Terms: conditions — Scleroderma, Systemic; Arthritis; Connective Tissue Diseases; Rare Diseases | interventions — Relaxin

INTERVENTIONS:
Drug: relaxin

SUMMARY:
OBJECTIVES: I. Determine whether parenteral relaxin improves skin tightness, Raynaud's phenomenon, digital morbidity, and digital ulcers in a patient with progressive systemic sclerosis (scleroderma).

II. Determine whether relaxin decreases collagen production by fibroblasts in vivo and cultured from skin biopsies.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a compassionate use study. The patient is treated with subcutaneous injections of recombinant relaxin for approximately 12 months. If clinically indicated, therapy may be extended.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Progressive systemic sclerosis (scleroderma)
* No pregnant or nursing women

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1
Dates: Start 1991-12; Study Completion 1997-12

CONTACTS AND LOCATIONS:
Overall Officials: G. Scott Herron, Study Chair — Stanford University